CLINICAL TRIAL: NCT02862457
Title: A Phase I Study of INCB024360 (Epacadostat) Alone, INCB024360 in Combination With Pembrolizumab (MK-3475), and INCB024360 and Pembrolizumab in Combination With Chemotherapy in Patients With Advanced Solid Tumors (KEYNOTE-434)
Brief Title: Study of Epacadostat (INCB024360) Alone and In Combination With Pembrolizumab (MK-3475) With Chemotherapy and Pembrolizumab Without Chemotherapy in Participants With Advanced Solid Tumors (MK-3475-434)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-434; MK-3475-434 (Other: Merck Protocol Number); 163423 (Registry Identifier: JAPIC-CTI)
Record Dates: First submitted 2016-08-03; First posted 2016-08-11 (Estimated); Results first posted 2022-01-11 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Neoplasms; Carcinoma, Non-Small-Cell Lung
Keywords: Advanced Solid Tumors; PD-1; PD1; Programmed Cell Death-1; Programmed Cell Death 1; Programmed Cell Death-Ligand 1 (PD-L1); Programmed Cell Death-Ligand 2 (PD-L2); PDL1; PDL2
MeSH Terms: conditions — Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — epacadostat; pembrolizumab; Cisplatin; Area Under Curve; Carboplatin; Pemetrexed; Paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Part A Cohort 1: epacadostat 25 mg (Experimental): Participants received 25 mg of epacadostat orally twice daily (BID) alone on Days 1-5 of Cycle 1 (28-day cycle) with a washout on Days 6 and 7. On Day 8 participants received a one-time intravenous (IV) infusion of 200 mg pembrolizumab while continuing to receive 25 mg of epacadostat BID on Days 8-28. For each 21-day cycle thereafter, participants received a one-time IV infusion of 200 mg pembrolizumab on Day 1 and received 25 mg of epacadostat BID on Days 1-21 for up to 35 cycles (approximately 2 years).
  Interventions: Drug: Epacadostat 25 mg; Biological: pembrolizumab 200 mg
- Part A Cohort 1: epacadostat 100 mg (Experimental): Participants received 100 mg of epacadostat orally BID alone on Days 1-5 of Cycle 1 (28-day cycle) with a washout on Days 6 and 7. On Day 8 participants received a one-time IV infusion of 200 mg pembrolizumab while continuing to receive 100 mg of epacadostat BID on Days 8-28. For each 21-day cycle thereafter, participants received a one-time IV infusion of 200 mg pembrolizumab on Day 1 and received 100 mg of epacadostat BID on Days 1-21 for up to 35 cycles (approximately 2 years).
  Interventions: Drug: Epacadostat 100 mg; Biological: pembrolizumab 200 mg
- Part A Cohort 2: epacadostat 25 mg+pembrolizumab (Experimental): For each 21-day cycle, participants received a one-time IV infusion of 200 mg pembrolizumab on Day 1 and received 25 mg of epacadostat orally BID on Days 1-21 for up to 35 cycles (approximately 2 years).
  Interventions: Drug: Epacadostat 25 mg; Biological: pembrolizumab 200 mg
- Part A Cohort 2: epacadostat 100 mg+pembrolizumab (Experimental): For each 21-day cycle, participants received a one-time IV infusion of 200 mg pembrolizumab on Day 1 and received 100 mg of epacadostat orally BID on Days 1-21 for up to 35 cycles (approximately 2 years).
  Interventions: Drug: Epacadostat 100 mg; Biological: pembrolizumab 200 mg
- Part B Cohort 1: pembrolizumab+cisplatin+pemetrexed (Experimental): For each 21-day cycle, participants received a one-time IV infusion of 200 mg pembrolizumab on Day 1 and 100 mg of epacadostat orally BID on Days 1-21 for up to 35 cycles (approximately 2 years). For the first 4 cycles, participants also received a one-time IV infusion of 75 mg/m^2 cisplatin and 500 mg/m^2 pemetrexed on Day 1. Treatment with epacadostat was stopped with protocol amendment 02.
  Interventions: Drug: Epacadostat 100 mg; Biological: pembrolizumab 200 mg; Drug: Cisplatin 75 mg/m^2; Drug: Pemetrexed 500 mg/m^2
- Part B Cohort 2: pembrolizumab+carboplatin+pemetrexed (Experimental): For each 21-day cycle, participants received a one-time IV infusion of 200 mg pembrolizumab on Day 1 and 100 mg of epacadostat orally BID on Days 1-21 for up to 35 cycles (approximately 2 years). For the first 4 cycles, participants also received a one-time IV infusion of Area Under the Curve (AUC) 5 carboplatin and 500 mg/m^2 pemetrexed on Day 1. Treatment with epacadostat was stopped with protocol amendment 02.
  Interventions: Drug: Epacadostat 100 mg; Biological: pembrolizumab 200 mg; Drug: Carboplatin Area Under the Curve (AUC) 5; Drug: Pemetrexed 500 mg/m^2
- Part B Cohort 3: pembrolizumab+carboplatin+paclitaxel (Experimental): For each 21-day cycle, participants received a one-time IV infusion of 200 mg pembrolizumab on Day 1 and 100 mg of epacadostat orally BID on Days 1-21 for up to 35 cycles (approximately 2 years). For the first 4 cycles, participants also received a one-time IV infusion of AUC 6 carboplatin and 200 mg/m^2 paclitaxel on Day 1. Treatment with epacadostat was stopped with protocol amendment 02.
  Interventions: Drug: Epacadostat 100 mg; Biological: pembrolizumab 200 mg; Drug: Paclitaxel 200 mg/m^2; Drug: Carboplatin AUC 6

INTERVENTIONS:
Drug: Epacadostat 25 mg — Oral administration
  Other Names: INCB024360
  Arms: Part A Cohort 1: epacadostat 25 mg; Part A Cohort 2: epacadostat 25 mg+pembrolizumab
Drug: Epacadostat 100 mg — Oral administration
  Other Names: INCB024360
  Arms: Part A Cohort 1: epacadostat 100 mg; Part A Cohort 2: epacadostat 100 mg+pembrolizumab; Part B Cohort 1: pembrolizumab+cisplatin+pemetrexed; Part B Cohort 2: pembrolizumab+carboplatin+pemetrexed; Part B Cohort 3: pembrolizumab+carboplatin+paclitaxel
Biological: pembrolizumab 200 mg — Intravenous (IV) infusion
  Other Names: MK-3475; KEYTRUDA®
Drug: Cisplatin 75 mg/m^2 — IV infusion
  Other Names: Platinol®; Platinol-AQ®
  Arms: Part B Cohort 1: pembrolizumab+cisplatin+pemetrexed
Drug: Carboplatin Area Under the Curve (AUC) 5 — IV infusion
  Other Names: Paraplatin®
  Arms: Part B Cohort 2: pembrolizumab+carboplatin+pemetrexed
Drug: Pemetrexed 500 mg/m^2 — IV infusion
  Other Names: Alimta®
  Arms: Part B Cohort 1: pembrolizumab+cisplatin+pemetrexed; Part B Cohort 2: pembrolizumab+carboplatin+pemetrexed
Drug: Paclitaxel 200 mg/m^2 — IV infusion
  Other Names: Taxol®; Abraxane®; Onxol®
  Arms: Part B Cohort 3: pembrolizumab+carboplatin+paclitaxel
Drug: Carboplatin AUC 6 — IV infusion
  Other Names: Paraplatin®
  Arms: Part B Cohort 3: pembrolizumab+carboplatin+paclitaxel

SUMMARY:
This is an open-label, non-randomized, Phase I study of epacadostat (INCB024360) alone and in combination with pembrolizumab with chemotherapy and pembrolizumab without chemotherapy in participants with advanced solid tumors. The primary objective of the trial is to evaluate the safety and tolerability of epacadostat administered alone and in combination with pembrolizumab with and without chemotherapy.

With protocol amendment 02 (26-April-2019), treatment with epacadostat was stopped in the "Epacad+Pembro+Cisplatin+Pemetrexed", "Epacad+Pembro+Carboplatin+Pemetrexed", and "Epacad+Pembro+Carboplatin+Paclitaxel" study arms.

ELIGIBILITY:
Inclusion Criteria:

* For Part A: Has a histologically-confirmed metastatic or locally advanced solid tumor that has failed to respond to standard therapy, progressed despite standard therapy, or for which standard therapy does not exist.
* For Part B: Has a histologically-confirmed or cytologically confirmed diagnosis of non-small cell lung carcinoma (NSCLC) stage IIIB/IV, be naïve to systemic therapy, and have confirmation that epidermal growth factor receptor (EGFR) or anaplastic lymphoma kinase (ALK)-directed therapy is not indicated. Cohort 1 and 2 must have a histological or cytological diagnosis of non-squamous cancer.
* Has at least one measurable lesion by computed tomography or magnetic resonance imaging per Response Evaluation Criteria In Solid Tumors (RECIST) 1.1
* Has Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Has a life expectancy of ≥3 months
* Females must not be pregnant (negative urine or serum human chorionic gonadotropin test within 72 hours of study start)
* Women of childbearing potential and male participants must agree to use adequate contraception during the study through 120 days after the last dose of study medication
* For Part A: Has provided tissue for programmed cell death ligand 1 (PD-L1)/ Indoleamine 2,3-dioxygenase 1 (IDO1) expression evaluation from an archival tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated. For Part B submission of tissue is optional.

Exclusion Criteria:

* Has received prior therapy with an anti-Programmed cell death protein (PD)-1, anti-PD-L1, anti-PD-L2, anti-CD137, anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) agents (including ipilimumab or any other antibody/drug specifically targeting T-cell co-stimulation or checkpoint pathways), or IDO1 inhibitor
* Is currently participating or has participated in a study with an investigational compound or device within 4 weeks, or 5 times half-life of the investigational compound, whichever is longer, of initial dosing on this study
* For Part A: Has had chemotherapy, targeted small molecule therapy, radiotherapy, major surgery, or biological cancer therapy (including monoclonal antibodies) within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to the first dose of study medication, or who has not recovered (≤ Grade 1 or baseline) from adverse events due to a previously administered treatment
* For Part B: Has received radiotherapy within 7 days of the first dose of trial treatment or radiation therapy to the lung that is >30 Gray (Gy) within 6 months of the first dose of study medication
* Is expected to require any other form of systemic or localized anti-neoplastic therapy while in study
* Has active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has symptomatic ascites or pleural effusion
* Has an active autoimmune disease that has required systemic treatment
* Is receiving systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 1 week prior to the first dose of study medication
* Has an active infection requiring systemic therapy
* Has history of (noninfectious) pneumonitis that required systemic steroids or current pneumonitis/interstitial lung disease
* Has received a live vaccine within 4 weeks prior to the first dose of study medication
* Has a known hypersensitivity to the components of the trial treatment or another monoclonal antibody
* For Part B: Has a known sensitivity to any component of cisplatin, carboplatin, paclitaxel, or pemetrexed.
* For Part B: Is on chronic systemic steroids with the exception of use of bronchodilators, inhaled steroids, or local steroid injections
* For Part B cohort 1 and 2: Is unable to interrupt aspirin or other nonsteroidal ant-inflammatory drugs (NSAIDs), other than an aspirin dose ≤1.3 g per day, for a 5-day period (8-day period for long-acting agents, such as piroxicam).
* For Part B cohort 1 and 2: Is unable or unwilling to take folic acid or vitamin B12 supplementation
* Is Human Immunodeficiency Virus (HIV)-positive (HIV 1/2 antibodies)
* Has known history of or is positive for active Hepatitis B (Hepatitis B surface antigen reactive) or has active Hepatitis C (Hepatitis C virus ribonucleic acid)
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children during the study through 120 days after the last dose of study medication
* Has received monoamine oxidase inhibitors (MAOIs) within the 3 weeks before the first dose of study medication
* Has any history of Serotonin Syndrome after receiving serotonergic drugs
* Has presence of a gastrointestinal condition that may affect drug absorption

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-08-23 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2020-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Yamamoto N, Satouchi M, Doi T, Fujiwara Y, Yanagitani N, Kawa Y, Yoh K, Leopold L, Munteanu M, Sawada T, Han S, Noguchi K, Nishio M. KEYNOTE-434 part B: A phase 1 study evaluating the combination of epacadostat, pembrolizumab, and chemotherapy in Japanese patients with previously untreated advanced non-small-cell lung cancer. Invest New Drugs. 2024 Jun;42(3):261-271. doi: 10.1007/s10637-024-01422-6. Epub 2024 Mar 26. PMID 38530565
- [Derived] Doi T, Fujiwara Y, Shitara K, Shimizu T, Yonemori K, Matsubara N, Ohno I, Kogawa T, Naito Y, Leopold L, Munteanu M, Yatsuzuka N, Han SR, Samkari A, Yamamoto N. The safety and tolerability of epacadostat alone and in combination with pembrolizumab in patients with advanced solid tumors: results from a first-in-Japanese phase I study (KEYNOTE-434). Invest New Drugs. 2021 Feb;39(1):152-162. doi: 10.1007/s10637-020-00942-1. Epub 2020 Jun 20. PMID 32564277

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Part A Cohort 1: Epacadostat 25 mg | Part A Cohort 1: Epacadostat 100 mg | Part A Cohort 2: Epacadostat 25 mg+Pembrolizumab | Part A Cohort 2: Epacadostat 100 mg+Pembrolizumab | Part B Cohort 1: Pembrolizumab+Cisplatin+Pemetrexed | Part B Cohort 2: Pembrolizumab+Carboplatin+Pemetrexed | Part B Cohort 3: Pembrolizumab+Carboplatin+Paclitaxel
Started | 3 | 3 | 3 | 6 | 7 | 6 | 6
Completed | 1 | 0 | 0 | 2 | 7 | 3 | 5
Not Completed | 2 | 3 | 3 | 4 | 0 | 3 | 1
Not completed — Death | 1 | 3 | 2 | 3 | 0 | 2 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population is all participants that received at least one dose of treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A Cohort 1: Epacadostat 25 mg | Part A Cohort 1: Epacadostat 100 mg | Part A Cohort 2: Epacadostat 25 mg+Pembrolizumab | Part A Cohort 2: Epacadostat 100 mg+Pembrolizumab | Part B Cohort 1: Pembrolizumab+Cisplatin+Pemetrexed | Part B Cohort 2: Pembrolizumab+Carboplatin+Pemetrexed | Part B Cohort 3: Pembrolizumab+Carboplatin+Paclitaxel | Total
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 7 | 6 | 6 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (7.8) | 71.0 (4.6) | 62.0 (12.2) | 67.5 (3.2) | 57.9 (7.3) | 68.0 (3.8) | 61.0 (13.4) | 63.9 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 1 | 1 | 3 | 1 | 12
  Male | 1 | 1 | 1 | 5 | 6 | 3 | 5 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 3 | 6 | 7 | 6 | 6 | 34
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 3 | 3 | 6 | 7 | 6 | 6 | 34
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Dose-Limiting Toxicities (DLTs) According to National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0 (NCI-CTCAE v.4.0)
Description: A DLT was defined as the occurrence of any treatment-emergent adverse event occurring up to and including Study Day 7 for Part A Cohort 1 or Day 21 for Part A Cohort 2 and Part B. The following criteria defined DLTs: Grade (G) 4 thrombocytopenia; G4 neutropenia (despite optimal supportive care in Part B) lasting >1 week; febrile neutropenia (only if considered clinically significant in Part B); G4 toxicity; G3 laboratory abnormality lasting >1 week: G3 toxicity excluding nausea or vomiting controlled within 72 hours, rash in the absence of desquamation, no mucosal involvement, does not require systemic steroids, and resolves to G1 by the next scheduled dose of pembrolizumab or 14 days; G2 or higher episcleritis, uveitis, or iritis; unable to receive 75% of epacadostat or 1 dose of pembrolizumab during the DLT observation period because of toxicity, even if the toxicity does not meet DLT criteria; or >2 week delay in initiating Cycle 2 due to toxicity.
Time Frame: Up to Day 7 for Part A Cohort 1; up to Day 21 for Part A Cohort 2 and Part B
Population: All participants in Parts A and B who received ≥1 dose of study treatment and who completed all safety evaluations in the pre-specified time frame for DLT analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Part A Cohort 1: Epacadostat 25 mg | Part A Cohort 1: Epacadostat 100 mg | Part A Cohort 2: Epacadostat 25 mg+Pembrolizumab | Part A Cohort 2: Epacadostat 100 mg+Pembrolizumab | Part B Cohort 1: Pembrolizumab+Cisplatin+Pemetrexed | Part B Cohort 2: Pembrolizumab+Carboplatin+Pemetrexed | Part B Cohort 3: Pembrolizumab+Carboplatin+Paclitaxel
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 7 | 6 | 6
Participants | 0 | 0 | 0 | 1 | 1 | 2 | 2

2. Primary Outcome: Number of Participants Who Experienced At Least One Adverse Event (AE)
Description: An adverse event is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An adverse event can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an adverse event. The number of participants who experienced an AE was reported for each arm.
Time Frame: Up to approximately 39.7 months
Population: All participants who received ≥1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A Cohort 1: Epacadostat 25 mg | Part A Cohort 1: Epacadostat 100 mg | Part A Cohort 2: Epacadostat 25 mg+Pembrolizumab | Part A Cohort 2: Epacadostat 100 mg+Pembrolizumab | Part B Cohort 1: Pembrolizumab+Cisplatin+Pemetrexed | Part B Cohort 2: Pembrolizumab+Carboplatin+Pemetrexed | Part B Cohort 3: Pembrolizumab+Carboplatin+Paclitaxel
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 7 | 6 | 6
Participants | 3 | 2 | 3 | 6 | 7 | 6 | 6

3. Primary Outcome: Number of Participants Who Discontinued Study Treatment Due to An Adverse Event (AE)
Description: An adverse event is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An adverse event can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an adverse event. The number of participants who discontinued due to an AE was reported for each arm.
Time Frame: Up to approximately 38.5 months
Population: All participants who received ≥1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A Cohort 1: Epacadostat 25 mg | Part A Cohort 1: Epacadostat 100 mg | Part A Cohort 2: Epacadostat 25 mg+Pembrolizumab | Part A Cohort 2: Epacadostat 100 mg+Pembrolizumab | Part B Cohort 1: Pembrolizumab+Cisplatin+Pemetrexed | Part B Cohort 2: Pembrolizumab+Carboplatin+Pemetrexed | Part B Cohort 3: Pembrolizumab+Carboplatin+Paclitaxel
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 7 | 6 | 6
Participants | 0 | 1 | 0 | 1 | 0 | 3 | 3

4. Secondary Outcome: Maximum Concentration (Cmax) of Epacadostat in Part A
Description: Cmax was the maximum observed concentration of epacadostat in plasma for epacadostat administered alone (Cohort 1) and epacadostat administered with pembrolizumab (Cohort 2). Per protocol, Cmax for Cohort 1 was measured on Days 1, 5, and 12 and Cmax for Cohort 2 was measured on Day 5 only. Blood samples were collected pre-dose and post-dose at multiple time points up to 12 days during Cycle 1 (28-day cycle). Cmax is presented as a geometric mean with a percent geometric coefficient of variation.
Time Frame: Cycle 1 (28-day cycle): Days 1, 5, and 12 at predose and 0.5, 1, 2, 4, 6, 8 and 10 hours postdose
Population: The analysis population consisted of all participants in Part A that contributed blood samples for analysis of Cmax. Per protocol, Cmax was only measured on Day 5 for Part A Cohort 2.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Part A Cohort 1: Epacadostat 25 mg | Part A Cohort 1: Epacadostat 100 mg | Part A Cohort 2: Epacadostat 25 mg+Pembrolizumab | Part A Cohort 2: Epacadostat 100 mg+Pembrolizumab
Number analyzed (Participants) | 3 | 3 | 3 | 6
nM
  Day 1: number analyzed (Participants) | 3 | 3 | 0 | 0
  Day 1 | 327 (15.9) | 1060 (19.7) |  |
  Day 5 | 269 (19.3) | 1100 (36.8) | 371 (10.7) | 852 (74.0)
  Day 12: number analyzed (Participants) | 3 | 3 | 0 | 0
  Day 12 | 294 (43.8) | 1200 (27.0) |  |

5. Secondary Outcome: Time to Maximum Concentration (Tmax) of Epacadostat in Part A
Description: Tmax was the time required to reach the maximum concentration of epacadostat in plasma for epacadostat administered alone (Cohort 1) and epacadostat administered with pembrolizumab (Cohort 2). Per protocol, Tmax for Cohort 1 was measured on Days 1, 5, and 12 and Tmax for Cohort 2 was measured on Day 5 only. Blood samples were collected pre-dose and post-dose at multiple time points up to 12 days during Cycle 1 (28-day cycle). Tmax is presented as a Median with a full range.
Time Frame: Cycle 1 (28-day cycle): Days 1, 5, and 12 at predose and 0.5, 1, 2, 4, 6, 8 and 10 hours postdose
Population: The analysis population consisted of all participants in Part A that contributed blood samples for analysis of Tmax. Per protocol, Tmax was only measured on Day 5 for Part A Cohort 2.
Measure: Median (Full Range); unit: hours
Arm/Group | Part A Cohort 1: Epacadostat 25 mg | Part A Cohort 1: Epacadostat 100 mg | Part A Cohort 2: Epacadostat 25 mg+Pembrolizumab | Part A Cohort 2: Epacadostat 100 mg+Pembrolizumab
Number analyzed (Participants) | 3 | 3 | 3 | 6
hours
  Day 1: number analyzed (Participants) | 3 | 3 | 0 | 0
  Day 1 | 2.00 [2.00 to 2.00] | 2.00 [2.00 to 2.00] |  |
  Day 5 | 2.00 [2.00 to 2.00] | 2.00 [2.00 to 4.00] | 2.00 [2.00 to 2.00] | 2.00 [1.00 to 4.00]
  Day 12: number analyzed (Participants) | 3 | 3 | 0 | 0
  Day 12 | 2.00 [2.00 to 2.00] | 2.00 [2.00 to 4.00] |  |

6. Secondary Outcome: Area Under the Concentration-Time Curve From Zero to the Time of the Last Measurable Concentration (AUC0-t) of Epacadostat in Part A
Description: AUC0-t was defined as the AUC from zero to the time of the last measurable concentration of epacadostat in plasma for epacadostat administered alone (Cohort 1) and epacadostat administered with pembrolizumab (Cohort 2). Per protocol, AUC0-t for Cohort 1 was measured on Days 1, 5, and 12 and AUC0-t for Cohort 2 was measured on Day 5 only. Blood samples were collected pre-dose and post-dose at multiple time points up to 12 days during Cycle 1 (28-day cycle). AUC0-t is presented as a geometric mean with a percent geometric coefficient of variation.
Time Frame: Cycle 1 (28-day cycle): Days 1, 5, and 12 at predose and 0.5, 1, 2, 4, 6, 8 and 10 hours postdose
Population: The analysis population consisted of all participants in Part A that contributed blood samples for analysis of AUC 0-t. Per protocol, AUC0-t was only measured on Day 5 for Part A Cohort 2.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM•hour
Arm/Group | Part A Cohort 1: Epacadostat 25 mg | Part A Cohort 1: Epacadostat 100 mg | Part A Cohort 2: Epacadostat 25 mg+Pembrolizumab | Part A Cohort 2: Epacadostat 100 mg+Pembrolizumab
Number analyzed (Participants) | 3 | 3 | 3 | 6
nM•hour
  Day 1: number analyzed (Participants) | 3 | 3 | 0 | 0
  Day 1 | 855 (13.0) | 4250 (7.1) |  |
  Day 5 | 1060 (24.0) | 4670 (22.7) | 1260 (8.8) | 3950 (38.8)
  Day 12: number analyzed (Participants) | 3 | 3 | 0 | 0
  Day 12 | 1020 (27.3) | 4710 (17.9) |  |

7. Secondary Outcome: Trough Concentration (Ctrough) of Epacadostat in Part A
Description: Ctrough was the lowest concentration of epacadostat in plasma just before the next dose for epacadostat administered alone (Cohort 1) and epacadostat administered with pembrolizumab (Cohort 2). Per protocol, Ctrough for Cohort 1 was measured on Days 1, 5, and 12 and Ctrough for Cohort 2 was measured on Day 5 only. Blood samples were collected pre-dose at multiple time points up to 12 days during Cycle 1 (28-day cycle). Ctrough is presented as a geometric mean with a percent geometric coefficient of variation.
Time Frame: Cycle 1 (28-day cycle): Days 1, 5, and 12 at predose
Population: The analysis population consisted of all participants in Part A that contributed blood samples for analysis of Ctrough. Per protocol, Ctrough was only measured on Day 5 for Part A Cohort 2.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Part A Cohort 1: Epacadostat 25 mg | Part A Cohort 1: Epacadostat 100 mg | Part A Cohort 2: Epacadostat 25 mg+Pembrolizumab | Part A Cohort 2: Epacadostat 100 mg+Pembrolizumab
Number analyzed (Participants) | 3 | 3 | 3 | 6
nM
  Day 1: number analyzed (Participants) | 3 | 3 | 0 | 0
  Day 1 | NA (NA) — Ctrough not calculated predose Cycle 1 Day 1 because it preceded exposure. | NA (NA) — Ctrough not calculated predose Cycle 1 Day 1 because it preceded exposure. |  |
  Day 5 | NA (NA) — Ctrough less than the limitation of quantification of the assay (20 nM). | 87.7 (21.7) | NA (NA) — Ctrough less than the limitation of quantification of the assay (20 nM). | 106.0 (64.1)
  Day 12: number analyzed (Participants) | 3 | 3 | 0 | 0
  Day 12 | NA (NA) — Ctrough less than the limitation of quantification of the assay (20 nM). | 95.4 (31.8) |  |

8. Secondary Outcome: Terminal Half-Life (t1/2) of Epacadostat in Part A
Description: t1/2 was the time required to divide the epacadostat concentration by two after reaching pseudo-equilibrium. Plasma t1/2 was measured for epacadostat administered alone (Cohort 1) and epacadostat administered with pembrolizumab (Cohort 2). Per protocol, t1/2 for Cohort 1 was measured on Days 1, 5, and 12 and t1/2 for Cohort 2 was measured on Day 5 only. Blood samples were collected pre-dose and post-dose at multiple time points up to 12 days during Cycle 1 (28-day cycle). t1/2 is presented as a geometric mean with a percent geometric coefficient of variation.
Time Frame: Cycle 1 (28-day cycle): Days 1, 5, and 12 at predose and 0.5, 1, 2, 4, 6, 8 and 10 hours postdose
Population: The analysis population consisted of all participants in Part A that contributed blood samples for analysis of t1/2. Per protocol, t1/2 was only measured on Day 5 for Part A Cohort 2.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part A Cohort 1: Epacadostat 25 mg | Part A Cohort 1: Epacadostat 100 mg | Part A Cohort 2: Epacadostat 25 mg+Pembrolizumab | Part A Cohort 2: Epacadostat 100 mg+Pembrolizumab
Number analyzed (Participants) | 3 | 3 | 3 | 6
hours
  Day 1: number analyzed (Participants) | 2 | 3 | 0 | 0
  Day 1 | 3.94 (NA) — Percent geometric coefficient of variation could not be calculated on data from 2 participants. | 2.55 (40.9) |  |
  Day 5 | 3.01 (70.6) | 2.82 (45.1) | 2.62 (9.7) | 3.77 (21.9)
  Day 12: number analyzed (Participants) | 3 | 3 | 0 | 0
  Day 12 | 4.27 (86.0) | 2.43 (16.1) |  |

9. Secondary Outcome: Maximum Concentration (Cmax) of Pembrolizumab in Part A Cycle 1
Description: Cmax was the maximum observed concentration of pembrolizumab in serum for participants that received either dose regimen in Part A for Cohort 1 combined, Cohort 2 combined, and Cohorts 1+2 combined. Per protocol, the analysis for the Cmax of pembrolizumab was performed in Cycle 1 only. Blood samples were collected predose and postdose within 30 minutes post pembrolizumab infusion during Cycle 1 (21-day pembrolizumab treatment cycle starting at Day 8 of Cycle 1). Cmax is presented as a geometric mean with a percent geometric coefficient of variation.
Time Frame: Cycle 1 (21-day pembrolizumab treatment cycle starting at Day 8 of Cycle 1): Day 1 predose and postdose within 30 minutes after the end of pembrolizumab infusion
Population: The analysis population consisted of all participants in Part A that contributed blood samples for analysis of Cmax. Per protocol, the Cmax of pembrolizumab for Part A was planned to be measured using data combined for Cohort 1 and Cohort 2 for the 200 mg pembrolizumab dose regimen irrespective of epacadostat dose received.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Groups:
- Part A Combined Cohort 1: All participants who received either dose (25 or 100 mg) of epacadostat orally twice daily (BID) alone on Days 1-5 of Cycle 1 (28-day cycle) with a washout on Days 6 and 7. On Day 8 participants received a one-time intravenous (IV) infusion of 200 mg pembrolizumab while continuing to receive 25 mg of epacadostat BID on Days 8-28. For each 21-day cycle thereafter, participants received a one-time IV infusion of 200 mg pembrolizumab on Day 1 and received either dose (25 or 100 mg) of epacadostat BID on Days 1-21.
- Part A Combined Cohort 2: All participants who received a one-time IV infusion of 200 mg pembrolizumab on Day 1 and received either dose (25 or 100 mg) of epacadostat orally BID on Days 1-21 for each 21-day cycle.
- Part A Combined Cohorts 1 and 2: All participants in Cohorts 1 and 2 combined.
Arm/Group | Part A Combined Cohort 1 | Part A Combined Cohort 2 | Part A Combined Cohorts 1 and 2
Number analyzed (Participants) | 6 | 9 | 15
µg/mL | 80.0 (12.3) | 73.8 (25.7) | 76.2 (21.1)

10. Secondary Outcome: Maximum Concentration (Cmax) of Pembrolizumab in Part B Cycle 1
Description: Cmax was the maximum observed concentration of pembrolizumab in serum for participants that received either dose regimen in Part B for Cohort 1, Cohort 2, Cohort 3, and Cohorts 1+2+ 3 combined. Per protocol, the analysis for the Cmax of pembrolizumab was performed in Cycle 1 only. Blood samples were collected predose and postdose within 30 minutes post pembrolizumab infusion during Cycle 1 (21-day pembrolizumab treatment cycle starting at Day 8 of Cycle 1). Cmax is presented as a geometric mean with a percent geometric coefficient of variation.
Time Frame: as for outcome 9
Population: The analysis population consisted of all participants in Part B that contributed blood samples for analysis of Cmax.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Groups:
- Part B Combined Cohorts 1, 2, and 3: All participants in Cohorts 1, 2, and 3 combined.
Arm/Group | Part B Cohort 1: Pembrolizumab+Cisplatin+Pemetrexed | Part B Cohort 2: Pembrolizumab+Carboplatin+Pemetrexed | Part B Cohort 3: Pembrolizumab+Carboplatin+Paclitaxel | Part B Combined Cohorts 1, 2, and 3
Number analyzed (Participants) | 7 | 6 | 6 | 19
µg/mL | 73.8 (25.0) | 64.3 (32.1) | 65.3 (22.4) | 68.0 (26.0)

11. Secondary Outcome: Trough Concentration (Ctrough) of Pembrolizumab in Part A Cycles 1, 2, 4, 6, and 8
Description: Ctrough was the lowest concentration of pembrolizumab in serum just before the next dose for participants that received either dose regimen in Part A for Cohort 1 combined, Cohort 2 combined, and Cohorts 1+2 combined. Per protocol, blood sampling for Ctrough was taken at predose prior to the Cycle 1, 2, 4, 6, and 8 infusion. Cycle 1 length was 28 days (21-day pembrolizumab treatment cycle starting at Day 8 of Cycle 1). Cycle 2, 4, 6, and 8 length was 21 days. Ctrough is presented as a geometric mean with a percent geometric coefficient of variation.
Time Frame: Predose prior to the Cycles 1, 2, 4, 6, and 8 infusion
Population: The analysis population consisted of all participants in Part A that contributed blood samples for analysis of Ctrough. Per protocol, the Ctrough of pembrolizumab for Part A was planned to be measured using data combined for Cohort 1 and Cohort 2 for the 200 mg pembrolizumab dose regimen irrespective of epacadostat dose received.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Part A Combined Cohort 1 | Part A Combined Cohort 2 | Part A Combined Cohorts 1 And 2
Number analyzed (Participants) | 6 | 9 | 15
µg/mL
  Cycle 1 | NA (NA) — Ctrough less than the limitation of quantification of the assay (20 nM) | NA (NA) — Ctrough less than the limitation of quantification of the assay (20 nM) | NA (NA) — Ctrough less than the limitation of quantification of the assay (20 nM)
  Cycle 2: number analyzed (Participants) | 6 | 8 | 14
  Cycle 2 | 17.3 (26.6) | 17.9 (33.5) | 17.6 (29.6)
  Cycle 4: number analyzed (Participants) | 3 | 6 | 9
  Cycle 4 | 24.5 (31.3) | 41.8 (21.1) | 35.0 (36.0)
  Cycle 6: number analyzed (Participants) | 3 | 4 | 7
  Cycle 6 | 28.5 (25.3) | 51.0 (17.4) | 39.8 (37.5)
  Cycle 8: number analyzed (Participants) | 1 | 3 | 4
  Cycle 8 | 38.2 (NA) — Percent geometric coefficient of variation could not be calculated on data from 1 participant. | 47.9 (13.9) | 45.2 (16.1)

12. Secondary Outcome: Trough Concentration (Ctrough) of Pembrolizumab in Part B Cycles 1, 2, 4, 6, and 8
Description: Ctrough was the lowest concentration of pembrolizumab in serum just before the next dose for participants that received either dose regimen in Part B for Cohort 1, Cohort 2, Cohort 3, and Cohorts 1+2+3 combined. Per protocol, blood sampling for Ctrough was taken at pre-dose prior to the Cycle 1, 2, 4, 6, and 8 infusion. Cycle 1 length was 28 days (21-day pembrolizumab treatment cycle starting at Day 8 of Cycle 1). Cycle 2, 4, 6, and 8 length was 21 days. Ctrough is presented as a geometric mean with a percent geometric coefficient of variation.
Time Frame: Predose prior to the Cycles 1, 2, 4, 6, and 8 infusion
Population: The analysis population consisted of all participants in Part B that contributed blood samples for analysis of Ctrough.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Part B Cohort 1: Pembrolizumab+Cisplatin+Pemetrexed | Part B Cohort 2: Pembrolizumab+Carboplatin+Pemetrexed | Part B Cohort 3: Pembrolizumab+Carboplatin+Paclitaxel | Part B Combined Cohorts 1, 2, and 3
Number analyzed (Participants) | 7 | 6 | 6 | 19
µg/mL
  Cycle 1 | NA (NA) — Ctrough less than the limitation of quantification of the assay (20 nM) | NA (NA) — Ctrough less than the limitation of quantification of the assay (20 nM) | NA (NA) — Ctrough less than the limitation of quantification of the assay (20 nM) | NA (NA) — Ctrough less than the limitation of quantification of the assay (20 nM)
  Cycle 2: number analyzed (Participants) | 6 | 3 | 5 | 14
  Cycle 2 | 16.6 (27.6) | 17.4 (36.6) | 8.69 (122) | 13.3 (73.9)
  Cycle 4: number analyzed (Participants) | 6 | 2 | 4 | 12
  Cycle 4 | 37.8 (20.2) | 28.1 (NA) — Percent geometric coefficient of variation could not be calculated on data from 2 participants. | 25.4 (25.7) | 31.5 (28.5)
  Cycle 6: number analyzed (Participants) | 5 | 2 | 3 | 10
  Cycle 6 | 53.8 (29.5) | 40.5 (NA) — Percent geometric coefficient of variation could not be calculated on data from 2 participants. | 21.5 (130) | 38.6 (73.5)
  Cycle 8: number analyzed (Participants) | 4 | 2 | 3 | 9
  Cycle 8 | 65.4 (18.6) | 52.7 (NA) — Percent geometric coefficient of variation could not be calculated on data from 2 participants. | 34.5 (42.9) | 50.3 (39.6)

ADVERSE EVENTS:
Time Frame: Up to approximately 39.7 months
Description: The analysis population for adverse events (AEs) and all-cause mortality consisted of all participants who received ≥1 dose of study treatment. Per protocol, disease progression was not considered an AE unless considered related to study treatment. Therefore, Medical Dictionary for Regulatory Activities (MedDRA) preferred terms neoplasm progression, malignant neoplasm progression, and disease progression not related to study treatment and/or did not result in death/hospitalization are excluded.
Arm/Group | Part A Cohort 1: Epacadostat 25 mg | Part A Cohort 1: Epacadostat 100 mg | Part A Cohort 2: Epacadostat 25 mg+Pembrolizumab | Part A Cohort 2: Epacadostat 100 mg+Pembrolizumab | Part B Cohort 1: Pembrolizumab+Cisplatin+Pemetrexed | Part B Cohort 2: Pembrolizumab+Carboplatin+Pemetrexed | Part B Cohort 3: Pembrolizumab+Carboplatin+Paclitaxel
All-Cause Mortality (participants affected / at risk) | 1/3 | 3/3 | 2/3 | 3/6 | 0/7 | 2/6 | 1/6
Serious Adverse Events (participants affected / at risk) | 0/3 | 2/3 | 2/3 | 1/6 | 1/7 | 2/6 | 2/6
Other Adverse Events (participants affected / at risk) | 3/3 | 2/3 | 3/3 | 6/6 | 7/7 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A Cohort 1: Epacadostat 25 mg (N=3) | Part A Cohort 1: Epacadostat 100 mg (N=3) | Part A Cohort 2: Epacadostat 25 mg+Pembrolizumab (N=3) | Part A Cohort 2: Epacadostat 100 mg+Pembrolizumab (N=6) | Part B Cohort 1: Pembrolizumab+Cisplatin+Pemetrexed (N=7) | Part B Cohort 2: Pembrolizumab+Carboplatin+Pemetrexed (N=6) | Part B Cohort 3: Pembrolizumab+Carboplatin+Paclitaxel (N=6)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cytomegalovirus colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A Cohort 1: Epacadostat 25 mg (N=3) | Part A Cohort 1: Epacadostat 100 mg (N=3) | Part A Cohort 2: Epacadostat 25 mg+Pembrolizumab (N=3) | Part A Cohort 2: Epacadostat 100 mg+Pembrolizumab (N=6) | Part B Cohort 1: Pembrolizumab+Cisplatin+Pemetrexed (N=7) | Part B Cohort 2: Pembrolizumab+Carboplatin+Pemetrexed (N=6) | Part B Cohort 3: Pembrolizumab+Carboplatin+Paclitaxel (N=6)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 3 (5) | 1 (2)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anal erosion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angular cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 6 (7) | 5 (5) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (5) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (8) | 5 (8) | 2 (6)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (2) | 2 (3) | 4 (4) | 2 (2) | 2 (3)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (2) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tracheitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Radiation skin injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 4 (9) | 2 (2) | 3 (6)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (4) | 2 (2) | 3 (5)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Blood thyroid stimulating hormone decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (9) | 2 (4) | 1 (4)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (9) | 1 (1) | 2 (5)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (6) | 2 (3)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 1 (4) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Vagus nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus genital (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail ridging (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (4) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 2 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vascular pain (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Vasculitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-26): https://cdn.clinicaltrials.gov/large-docs/57/NCT02862457/Prot_SAP_000.pdf